CLINICAL TRIAL: NCT00225836
Title: Treatment of Dysmenorrhoea With the OVA TENS Apparatus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Vitacon AS, Vegamot 8, 7048 Trondheim, Norway (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OVA study
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Dysmenorrhoea
Keywords: Dysmenorrhoea; Women; Pain; TENS
MeSH Terms: conditions — Dysmenorrhea; Pain

INTERVENTIONS:
Device: OVA (TENS apparatus)

SUMMARY:
Dysmenorrhoea (menstrual pain) is a common complaint among women, leading to use of analgesics, reduced quality of life, and interference with daily activities such as going to work or school.

Transcutaneous electrical nerve stimulation (TENS) is a well established method for treatment of pain. Several clinical studies have shown TENS treatment to be effective against dysmenorrhoea. A TENS apparatus specifically developed for the treatment of dysmenorrhoea has now become commercially available (OVA), but is has not been tested in clinical studies.

This study will be done to evaluate the clinical utility of treatment with OVA in women with primary dysmenorrhoea.

DETAILED DESCRIPTION:
Study aims: To compare perception of dysmenorrhoea with and without use of OVA.

Design: Prospective, clinical study lasting four months. The women will use the OVA apparatus during every other menstruation.

Inclusion: 20 female volunteers with primary dysmenorrhoea.

Exclusion: Pregnancy, either ongoing or planned during the study period. Secondary dysmenorrhoea.

Consent: The participants will receive verbal and written information and will sign a consent form.

Randomisation: The participants are randomised to start with either active treatment or observation by drawing a closed, opaque envelope containing the forms for registration of perception of pain.

Registering pain: The participants will mark their perceived degree of dysmenorrhoea daily on 10 cm visual analogue scale (VAS) during each menstruation.

Filling in forms: During each of the four menstruations throughout the study period the participants will respond daily to the questions on the form and note degree of pain on the VAS. At the end of each menstruation they will mail the current form in a stamped and addressed envelope to the study coordinator.

Statistics: We assume that a difference of 2 VAS-points is required for an effect to be of clinical interest. One-sided t-test for paired data will be used in the analysis.

Power calculation using the statistics program SSD v7.0 has shown that 16 participants is required to demonstrate a difference of 2 points at level of significance p=0.01, 90% power and assumed standard deviation of 2.

ELIGIBILITY:
Inclusion Criteria:

* Primary dysmenorrhoea

Exclusion Criteria:

* Pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Change in VAS pain score

CONTACTS AND LOCATIONS:
Overall Officials: Hjalmar A Schiotz, MD, PhD, Principal Investigator — Consultant Gynecologist, The Hospital of Vestfold, Tonsberg, Norway
Locations (1):
- Dept of Ob/Gyn, The Hospital of Vestfold, Tønsberg, Norway